CLINICAL TRIAL: NCT00204334
Title: Effects of Anemia Correction on Vascular Function, Endothelial Cell Markers and Monocyte Apoptosis in Renal Transplant Recipients
Brief Title: Effects of Anemia Correction on Vascular and Monocyte Function in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Amgen (Industry)
Responsible Party: University Hospital Muenster, University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Haus_Lang-Endothel-Mono-Hb; DE-2004-4077
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-05

CONDITIONS: Kidney Transplantation; Anemia
Keywords: Kidney transplantation; anemia; vascular endothelium; monocytes; apoptosis
MeSH Terms: conditions — Anemia

INTERVENTIONS:
Drug: darbopoeitin

SUMMARY:
Correction of anaemia in renal transplant recipients by parenteral application of recombinant erythropoietin and if necessary iron will improve large artery function (endothelial function and elasticity), as assessed by ultrasound techniques and applanation tonometry.

The changes in large artery function will be reflected by changes in serological markers of endothelial function and oxidative stress and by changes in monocyte function and apoptosis.

There are gender differences in the responses of vascular function to correction of anemia.

Besides improvement of large artery function, correction of anemia will also affect parameters of graft function, i.e. glomerular and tubular proteinuria.

DETAILED DESCRIPTION:
The value of anaemia therapy with recombinant erythropoietin and iron for improvement of cardiovascular outcome has been clearly demonstrated in dialysis patients and is standard of care. In this patient collective one study shows that correction of anaemia together with blood pressure control does improve large artery function. After kidney transplantation, the situation is not clear. Anemia is common in kidney transplant patients despite a functioning graft and is caused by inadequate erythropoietin production, inflammatory reactions and toxic bone marrow depression. Current guidelines suggest to correct anemia also in kidney transplant recipients in analogy to hemodialysis patients, however, there is to date no evidence that correction of mild to moderate anemia will improve cardiovascular outcome. Since cardiovascular outcome studies are difficult to perform in renal transplant patients we propose to study intermediate endpoints, surrogate parameters of cardiovascular endpoints, i.e. large artery distensibility and endothelium-dependent brachial artery dilatation. Our group was able to show that the former is a valid marker of cardiovascular morbidity in renal transplant patients (1), and a recent report stated the same prognostic value for brachial artery flow-dependent dilatation in hemodialysis patients. Since the causes of anemia in renal transplant patients are complex, it is not clear that treatment of at anemia with recombinant erythropoietin and iron will be beneficial. Erythropoetin treatment is likely to improve hypoxia and thereby to improve large artery function, but also upregulates circulating endothelial progenitor cells, already elevated in kidney transplant patients and a marker of vascular stress, e.g. in patients with vasculitis. Erythropoietin might therefore be detrimental to endothelial function and as a consequence to vascular elasticity. It may be argued that in renal transplant patients, vascular damage is profound and irreversible and therefore vascular function does not respond to pharmacological interventions. However, our group was able to show that although renal transplant patients have severely impaired large artery functional wall properties independent of immunosuppressive treatment regimens (2), they have a preserved large artery vasodilator capacity (3) and that treatment with a statin produces sustained long-term improvements of endothelial function in kidney transplant patients (4). Previous studies showed effects of erythropoietin treatment on serological parameters of endothelial function in hemodialysis patients. It is important to relate erythropoietin-induced changes in these parameters to changes in large artery function. Particularly, in the aimed target population immunological processes are very likely to affect vascular function. It has been shown that endothelial cell proliferation is induced by angiogenetic factors released by activated monocytes. Besides monocyte adhesion to endothelial cells is triggered e.g. by endothelial cells themselves when they are exposed to shear stress(5). During the adhesion process different costimulatory factors become important in the early and critical atherogenetic event. Monocyte survival and activation do have a key role in this process leading to arteriosclerosis and endothelial damage(6). Changes in monocyte survival in dependence of immunosuppression or erythropoietin treatment may be responsible for increasing circulating endothelial cells(7). Therefore we aim to relate erythropoietin-induced changes in vascular function to changes in monocyte function and apoptosis. In many disease states changes in endothelial function are reflected by changes in urinary protein excretion. Therefore, erythropoietin therapy could alter urinary protein excretion in parallel to the changes observed in large artery function. Finally, anemia is more common in female renal transplant recipients than in male renal transplant recipients, and female dialysis patients tend to require more erythropoietin for anemia treatment that male patients. Therefore it is conceivable that gender differences exist with respect to the effects of anemia correction on vascular function.

1. Barenbrock, M., M. Kosch, E. Joster, K. Kisters, K. H. Rahn, and M. Hausberg. Reduced arterial distensibility is a predictor of cardiovascular disease in patients after renal transplantation. J.Hypertens. 2002, 20: 79-84
2. Kosch M, Hausberg M, Suwelack B. Studies on effects of calcineurin inhibitor withdrawal on arterial distensibility and endothelial function in renal transplant recipient. Transplantation 2003, 76:1516-9.
3. Hausberg M, Kisters K, Kosch M, Rahn KH, Barenbrock M. Flow-mediated vasodilation and distensibility of the brachial artery in renal allograft recipients. Kidney Int 1999, 55: 1104-1110
4. Kosch M, Barenbrock M, Suwelack B, Schaefer RM, Rahn KH, Hausberg M. Effect of a 3-year therapy with the 3-hydroxy-3-methylglutaryl coenzyme a reductase-inhibitor fluvastatin on endothelial function and distensibility of large arteries in hypercholesterolemic renal transplant recipient. Am J Kidney Dis. 2003, 41:1088-96
5. Hwang J, Saha A, Boo YC, Sorescu GP, McNally JS, Holland SM, Dikalov S, Giddens DP, Griendling KK, Harrison DG, Jo H. Oscillatory shear stress stimulates endothelial production of O2- from p47phox-dependent NAD(P)H oxidases, leading to monocyte adhesion. J Biol Chem. 2003,278(47): 47291-47298.
6. Österud A, Björklid E. Role of monocytes in atherogenesis. Physiological reviews, 2003, 83: 1069-1112.
7. Bahlmann FH, DeGroot K, Duckert T, Niemczyk E, Bahlmann E, Boehm SM, Haller H, Fliser D. Endothelial progenitor cell proliferation and differentiation is regulated by erythropoietin. Kidney Int. 2003; 64:1648-1652.

ELIGIBILITY:
Inclusion Criteria:

kidney transplant recipient stable kidney function Hb between 10mg/ml and 10.5mg/ml

Exclusion Criteria:

acute rejection Hb above 12.0mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Vessel wall stiffness

SECONDARY OUTCOMES:
expression of endothelial cell markers

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hausberg, MD, Principal Investigator — UKM- Medical Department D
Locations (1):
- UKM, Münster, North Rhine-Westphalia, Germany